CLINICAL TRIAL: NCT04651933
Title: A Training Set for the Homologous Recombination Deficiency Scoring Model With Loss of Heterozygosity Status in Epithelial Ovarian Cancer
Brief Title: A Training Set for the HRD Model in EOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-LOH
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Epithelial Ovarian Cancer; BRCA Mutation; Loss of Heterozygosity; Prognosis; Platinum Resistance; Homologous Recombination Deficiency
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples from the patients' peripheral blood and tumor tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epithelial ovarian cancer patients sensitive to platinum based chemotherapy
  Interventions: Genetic: Homologous recombination deficiency model
- Epithelial ovarian cancer patients resistant to platinum based chemotherapy
  Interventions: Genetic: Homologous recombination deficiency model

INTERVENTIONS:
Genetic: Homologous recombination deficiency model — A homologous recombination deficiency (HRD) scoring model based on loss of heterozygosity (LOH)

SUMMARY:
A homologous recombination deficiency (HRD) scoring model based on loss of heterozygosity (LOH) is little explored in epithelial ovarian cancer (EOC) patients. This study would recruit 200 Chinese EOC patients with known BRCA1/2 mutation status and resistance to platinum-based chemotherapy. A LOH-HRD model is to be constructed based on the genetic testing in these patients. The mutated genes, HRD score model and their relationship with the prognosis, would provide a full description of for the Chinese EOC patients, and a potential explanation of platinum-resistance in such population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathological confirmation of epithelial ovarian cancer
* With available tumor tissues
* Given consents to participate the study

Exclusion Criteria:

• Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known BRCA1/2 mutation status and resistance to platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2022-11-26 (Estimated)

PRIMARY OUTCOMES:
Homologous recombination deficiency (HRD) score | Two years
  The HRD score for individual patient is a scale describing her HRD status. The score model is calculated by the analysis for loss of heterozygosity (LOH), and the minimum value is 0, but the maximun value is not available. Higher scores mean more sensitivity to poly-ADP-ribose polymerase inhibitor

SECONDARY OUTCOMES:
Progression-free survival | Five years
  Progression-free survival in recruited patients
Overall survival | Five years
  Overall survival in recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China